CLINICAL TRIAL: NCT00811018
Title: A Long-Term, Open-Label Study To Evaluate The Safety Of Sitaxsentan Sodium Treatment In Patients With Pulmonary Arterial Hypertension
Acronym: STRIDE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This trial was prematurely terminated on Dec 9 2010 due to safety concerns, specifically emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: B1321007; FPH03
Record Dates: First submitted 2008-12-09; First posted 2008-12-18 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2011-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Open-label study
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — sitaxsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitaxsentan (Experimental): Sitaxsentan
  Interventions: Drug: Sitaxsentan

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan 100 mg tablets once daily
  Other Names: Sitaxentan

SUMMARY:
This is a multi-center, open-label study of sitaxsentan sodium 100 mg taken orally once daily by subjects with PAH until sitaxsentan, in a particular country or region, is commercially available for the treatment of PAH or the study is closed.

DETAILED DESCRIPTION:
Open-label extension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pulmonary Arterial Hypertension (PAH) confirmed by cardiac catheterization.
* Current diagnosis of WHO group 1 PAH with functional class 2, 3, or 4 symptoms.

Exclusion Criteria:

* Has portal hypertension or chronic liver disease.
* Has history of left sided heart disease or significant cardiac disease.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1192 (Actual)
Dates: Start 2003-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- United States (34):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Torrence, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Capital Federal
- Australia (4):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Chermside Q, Queensland
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, Chermside
- Austria (2):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Vienna
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Brazil (3):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo
- Canada (7):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- France (3):
  - Pfizer Investigational Site, Clamart
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Strasbourg
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Giessen
  - Pfizer Investigational Site, Greifswald
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Regensburg
- Israel (2):
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel-Hashomer, Ramat Gan
- Pfizer Investigational Site, Bologna, Italy
- Mexico (3):
  - Pfizer Investigational Site, Monterrey, CP
  - Pfizer Investigational Site, Tlalpan, Mexico City
  - Pfizer Investigational Site, Monterrey, N.l.
- Pfizer Investigational Site, Amsterdam, Netherlands
- Poland (3):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze
- Pfizer Investigational Site, Barcelona, Barcelona, Spain
- United Kingdom (4):
  - Pfizer Investigational Site, Papworth Everard, Cambridgeshire
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321007&StudyName=A%20Long-Term%2C%20Open-Label%20Study%20to%20Evaluate%20the%20Safety%20of%20Sitaxsentan%20Sodium%20Treatment%20in%20Patients%20with%20Pulmonary%20Arterial%20Hypertension

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from studies FPH02/FPH02-X (STRIDE 2/STRIDE 2 Extension [NCT00080457, NCT00593905]), FPH04 (STRIDE 4), FPH06 (STRIDE 6) or were naive to sitaxsentan sodium.
Groups:
- Sitaxsentan: All participants received sitaxsentan 100 milligrams (mg) orally once daily beginning on Study Day 1 to termination from study.
Period: Overall Study
Arm/Group | Sitaxsentan
Started | 1192
Completed | 224
Not Completed | 968
Not completed — Additional Chronic Treatment | 31
Not completed — Adverse Event | 79
Not completed — Death | 147
Not completed — ALT/AST >3x UNL, Bilirubin >2xUNL | 4
Not completed — ALT/AST >5x Upper Limit of Normal (ULN) | 70
Not completed — Investigator Decision | 57
Not completed — Lost to Follow-up | 19
Not completed — Pregnancy | 6
Not completed — Sponsor Decision | 450
Not completed — Withdrawal by Subject | 70
Not completed — WHO FC deterioration and 6MWD decrease | 9
Not completed — Other | 26

BASELINE CHARACTERISTICS:
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
Age, Customized [Number; unit: participants]
  less than (<) 18 years | 35
  18-44 years | 433
  45-64 years | 468
  greater than or equal to 65 years | 256
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 914
  Male | 278

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product were reported.
Time Frame: Day 1 up to 82 months
Population: Safety Population: all enrolled participants who took at least one dose of sitaxsentan 100 mg during the study
Measure: Number; unit: participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
participants
  AEs | 1150
  SAEs | 586

2. Primary Outcome: The Percentage of Participants Who Experience an Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) Value Greater Than (>) 3.0 Times (x) the Upper Limit of Normal Range (ULN)
Description: ALT and AST data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 62, 68, 72, 74, 80, 84, 88, 92, 96, 100, 104, 108 and every 4 weeks to Termination up to 82 months
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
percentage of participants
  > 3 x ULN and less than or equal to (<=) 5x ULN | 5.12
  > 5 x ULN and <= 8 x ULN | 4.45
  > 8 x ULN and <= 10 x ULN | 0.76
  > 10 x ULN | 2.60

3. Primary Outcome: The Percentage of Participants Who Experience an ALT and AST Value > 3.0 x ULN
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
percentage of participants
  > 3 x ULN and <= 5 x ULN | 3.94
  > 5 x ULN and <= 8 x ULN | 2.60
  > 8 x ULN and <= 10 x ULN | 0.67
  > 10 x ULN | 1.26

4. Primary Outcome: Percentage of Participants With Total Bilirubin > 1.5 x ULN
Description: Total builirubin data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: as for outcome 2
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
percentage of participants
  >= 1.5 x ULN and <2 x ULN | 10.23
  >= 2 x ULN and < 3x ULN | 6.80
  >= 3x ULN | 5.03

5. Primary Outcome: Percentage of Participants With Laboratory Test Abnormalities (Hematology)
Description: Hematology data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: as for outcome 2
Population: Safety Population; N=number of participants with normal observation at baseline; n=number of participants with normal baseline and an abnormality meeting specific criteria for the specific lab
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 814
percentage of participants
  Basophiles (n=814) | 4.1
  Eosinophiles % (n=3) | 100
  Eosinophils (n=785) | 20.6
  Hematocrit (n=537) | 46.2
  Hemoglobin (n=573) | 48.7
  Lymphocytes (n=737) | 35.5
  Mean Corpuscular Hemoglobin (n=56) | 21.4
  Mean Corpuscular Hemoglobin Concentration (n=59) | 33.9
  Mean Corpuscular Volume (n=65) | 27.7
  Monocytes (n=766) | 28.3
  Neutrophiles (n=728) | 38
  Platelets Count (n=719) | 26.3
  Red Blood Cells (n=542) | 39.1
  White Blood Cells (n=730) | 35.3

6. Primary Outcome: Percentage of Participants With Laboratory Test Abnormalities (Chemistry)
Description: Chemistry data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 839
percentage of participants
  Albumin (n=33) | 45.5
  Alkaline Phosphatase (n=593) | 45.5
  ALT (n=839) | 36.1
  Amylase (n=9) | 0
  AST (n=814) | 49.4
  Bicarbonate (n=540) | 56.7
  Blood urea nitrogen (BUN) (n=615) | 42.4
  Calcium (n=819) | 21.4
  Chloride (n=804) | 31
  Creatinine (n=808) | 25
  Direct Bilirubin (n=11) | 54.5
  Gamma glutamyltransferase (GGT) (n=22) | 45.5
  Glucose (n=674) | 61.6
  Glucose-fasting (n=2) | 50
  Indirect Bilirubin (n=11) | 45.5
  Phosphorus (n=740) | 50.8
  Potassium (n=749) | 51.8
  Sodium (n=811) | 29.1
  Total Bilirubin (n=726) | 27.7
  Total Protein (n=738) | 38.1
  Urea (n=35) | 48.6
  Uric Acid (n=415) | 46.5

7. Primary Outcome: Percentage of Participants With Laboratory Test Abnormalities (Urinalysis)
Description: Urinalysis data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 789
percentage of participants
  PH (n=789) | 0
  Specific Gravity (n=787) | 1.8

8. Primary Outcome: Percentage of Participants With Anticoagulant Use
Description: Participants with anticoagulant use before first dose or participants with anticoagulant use from first dose of sitaxsentan.
Time Frame: Baseline, Weeks 1 and 2, every 2 weeks up to Week 52, Amendment 4 visit, every 4 weeks up to 82 months
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
percentage of participants
  Warfarin before first dose | 39.77
  Warfarin Derivatives before first dose | 19.13
  Other Anticoagulants before first dose | 2.01
  Warfarin from first dose/data cut off | 58.22
  Warfarin Derivatives from first dose/data cut off | 20.55
  Other Anticoagulants from first dose/data cut off | 2.52

9. Primary Outcome: Percentage of Participants With Elevated International Normalize Ratio (INR)
Description: Elevated INR in participants who took warfarin, warfarin derivatives, other anticoagulant and no anticoagulants. Elevated INR defined as > 3.5. Percentage calculated using number of participants with INR data as the denominator.
Time Frame: Baseline, Weeks 1 and 2, every 2 weeks up to Week 52, Amendment 4 visit, every 4 weeks up to 82 months
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 1192
percentage of participants
  INR <= 3.5; warfarin | 20.97
  INR >3.5 and <=5; warfarin | 17.70
  INR >5 and <=9; warfarin | 12.75
  INR > 9; warfarin | 3.44
  INR <=3.5; warfarin derivatives | 4.95
  INR >3.5 and <=5; warfarin derivatives | 6.96
  INR >5 and <=9; warfarin derivatives | 5.96
  INR >9; warfarin derivatives | 1.85
  INR <=3.5; other anticoagulant | 1.34
  INR >3.5 and <=5; other anticoagulant | 0.59
  INR >5 and <= 9; other anticoagulant | 0.50
  INR <=3.5; no anticoagulant | 19.55
  INR >3.5 and <= 5; no anticoagulant | 0.17
  INR >5 and <=9; no anticoagulant | 0.42
  INR >9; no anticoagulant | 0.25

10. Primary Outcome: Percentage of Participants With Electrocardiography (ECG) Results of Potential Clinical Importance
Description: Standard 12-lead ECG results determined to be of potential clinical importance according to investigator clinical judgement.
Time Frame: Weeks 28,60,72,84,96,104, Transition Visit up to 82 months
Population: Data not summarized, study terminated early
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 0

11. Primary Outcome: Percentage of Participants With Vital Sign Results of Potential Clinical Importance
Description: Vital signs include sitting blood pressure, respiration rate, heart rate and temperature. Potential clinical importance determined according to investigator clinical judgement.
Time Frame: Day 1, Weeks 28,60,72,84,96,104, Transition visit, every 6 months Post Transition, up to 82 months
Population: Data not summarized, study terminated early
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 0

12. Primary Outcome: Percentage of Participants With Abnormal Prothrombin Time (PT)
Description: PT data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: Baseline, Weeks 1 and 2, every 2 weeks up to Week 52, Amendment 4 visit, every 4 weeks up to 82 months
Population: Data not summarized, study terminated early
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 0

13. Primary Outcome: Percentage of Participants With Abnormal Partial Thromboplastin Time (PTT)
Description: PTT data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analysis.
Time Frame: Baseline, Weeks 1 and 2, every 2 weeks up to Week 52, Amendment 4 visit, every 4 weeks up to 82 months
Population: Data not summarized, study terminated early
Measure: Number; unit: percentage of participants
Arm/Group | Sitaxsentan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan
Serious Adverse Events (participants affected / at risk) | 586/1192
Other Adverse Events (participants affected / at risk) | 1069/1192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=1192)
Anaemia (Blood and lymphatic system disorders) | 16
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 16
Atrial flutter (Cardiac disorders) | 15
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 5
Cardiac aneurysm (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 8
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 26
Cardiac failure congestive (Cardiac disorders) | 14
Cardiac pseudoaneurysm (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 5
Cor pulmonale (Cardiac disorders) | 7
Cor pulmonale acute (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Low cardiac output syndrome (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 9
Myocardial ischaemia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 6
Right atrial dilatation (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 68
Sick sinus syndrome (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 7
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 2
Ventricular dysfunction (Cardiac disorders) | 3
Ventricular failure (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 3
Ventricular tachycardia (Cardiac disorders) | 3
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Blindness (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Abdominal haematoma (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 1
Appendix disorder (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 4
Large intestine perforation (Gastrointestinal disorders) | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Oesophageal disorder (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 2
Pancreatic mass (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Volvulus (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 5
Cardiac death (General disorders) | 1
Catheter related complication (General disorders) | 2
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 25
Condition aggravated (General disorders) | 1
Death (General disorders) | 3
Device dislocation (General disorders) | 2
Fatigue (General disorders) | 3
Generalised oedema (General disorders) | 2
Hyperpyrexia (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Mass (General disorders) | 1
Medical device complication (General disorders) | 1
Multi-organ failure (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 6
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 17
Systemic inflammatory response syndrome (General disorders) | 2
Therapeutic response unexpected (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 8
Cholecystitis acute (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Abdominal infection (Infections and infestations) | 1
Abdominal sepsis (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 5
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 12
Bronchitis acute (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 5
Campylobacter infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 5
Catheter sepsis (Infections and infestations) | 4
Catheter site infection (Infections and infestations) | 6
Cellulitis (Infections and infestations) | 5
Central line infection (Infections and infestations) | 4
Chronic sinusitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Dermo-hypodermitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 4
Diarrhoea infectious (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 3
Escherichia bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Mycobacterial infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Peritonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 65
Pneumonia klebsiella (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 1
Pyometra (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 4
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 2
Viral pericarditis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Chest injury (Injury, poisoning and procedural complications) | 1
Collapse of lung (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 5
Tibia fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Angiogram (Investigations) | 1
Apnoea test (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Aspiration bronchial (Investigations) | 1
Biopsy (Investigations) | 1
Biopsy lung (Investigations) | 1
Bleeding time prolonged (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Bronchoscopy (Investigations) | 1
Catheterisation cardiac (Investigations) | 14
Catheterisation cardiac normal (Investigations) | 1
Diagnostic procedure (Investigations) | 1
ECG signs of myocardial ischaemia (Investigations) | 1
Echocardiogram abnormal (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Heart rate increased (Investigations) | 1
Hepatic enzyme abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 3
International normalised ratio increased (Investigations) | 6
Intraocular pressure increased (Investigations) | 1
Investigation (Investigations) | 2
Liver function test abnormal (Investigations) | 5
Oxygen consumption increased (Investigations) | 1
Physical examination (Investigations) | 5
Pregnancy test positive (Investigations) | 1
Troponin increased (Investigations) | 1
Volume blood increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Electrolyte depletion (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 10
Fluid retention (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperosmolar state (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 7
Hypovolaemia (Metabolism and nutrition disorders) | 1
Articular calcification (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
CREST syndrome (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral hypoperfusion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 4
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Embolic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Ischaemic stroke (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 23
Transient ischaemic attack (Nervous system disorders) | 5
Vocal cord paralysis (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Missed labour (Pregnancy, puerperium and perinatal conditions) | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Acute stress disorder (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Schizoaffective disorder (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 10
Renal failure chronic (Renal and urinary disorders) | 2
Ureteric haemorrhage (Renal and urinary disorders) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Reproductive tract disorder (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 71
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 62
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Anticoagulant therapy (Surgical and medical procedures) | 1
Appendicectomy (Surgical and medical procedures) | 1
Arterial stent insertion (Surgical and medical procedures) | 1
Atrial septal defect repair (Surgical and medical procedures) | 3
Balloon atrial septostomy (Surgical and medical procedures) | 1
Cardiac ablation (Surgical and medical procedures) | 2
Cardiac operation (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Cardioversion (Surgical and medical procedures) | 2
Catheter placement (Surgical and medical procedures) | 2
Central venous catheter removal (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Cholelithotomy (Surgical and medical procedures) | 1
Colostomy closure (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Drug therapy (Surgical and medical procedures) | 13
Endarterectomy (Surgical and medical procedures) | 1
Endotracheal intubation (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Foot amputation (Surgical and medical procedures) | 1
Heart and lung transplant (Surgical and medical procedures) | 3
Hernia diaphragmatic repair (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 3
Hysterectomy (Surgical and medical procedures) | 1
Infusion (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Intraocular lens implant (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Lens implant (Surgical and medical procedures) | 1
Lung transplant (Surgical and medical procedures) | 1
Lymphadenectomy (Surgical and medical procedures) | 1
Office visit (Surgical and medical procedures) | 3
Packed red blood cell transfusion (Surgical and medical procedures) | 1
Pain management (Surgical and medical procedures) | 1
Phlebectomy (Surgical and medical procedures) | 1
Prophylaxis against gastrointestinal ulcer (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Routine health maintenance (Surgical and medical procedures) | 2
Spinal cord operation (Surgical and medical procedures) | 1
Spinal decompression (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 3
Therapy cessation (Surgical and medical procedures) | 1
Therapy regimen changed (Surgical and medical procedures) | 1
Toe amputation (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Transplant (Surgical and medical procedures) | 1
Transurethral bladder resection (Surgical and medical procedures) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Vascular bypass graft (Surgical and medical procedures) | 1
Wound treatment (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 4
Hyperaemia (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 10
Hypovolaemic shock (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=1192)
Anaemia (Blood and lymphatic system disorders) | 77
Palpitations (Cardiac disorders) | 137
Abdominal pain (Gastrointestinal disorders) | 93
Abdominal pain upper (Gastrointestinal disorders) | 80
Constipation (Gastrointestinal disorders) | 82
Diarrhoea (Gastrointestinal disorders) | 211
Nausea (Gastrointestinal disorders) | 228
Vomiting (Gastrointestinal disorders) | 104
Chest pain (General disorders) | 201
Fatigue (General disorders) | 224
Oedema (General disorders) | 83
Oedema peripheral (General disorders) | 287
Bronchitis (Infections and infestations) | 100
Influenza (Infections and infestations) | 67
Nasopharyngitis (Infections and infestations) | 219
Sinusitis (Infections and infestations) | 115
Upper respiratory tract infection (Infections and infestations) | 306
Urinary tract infection (Infections and infestations) | 115
Aspartate aminotransferase increased (Investigations) | 68
International normalised ratio increased (Investigations) | 157
Liver function test abnormal (Investigations) | 79
Hypokalaemia (Metabolism and nutrition disorders) | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 134
Back pain (Musculoskeletal and connective tissue disorders) | 137
Muscle spasms (Musculoskeletal and connective tissue disorders) | 74
Pain in extremity (Musculoskeletal and connective tissue disorders) | 163
Dizziness (Nervous system disorders) | 243
Headache (Nervous system disorders) | 294
Syncope (Nervous system disorders) | 76
Anxiety (Psychiatric disorders) | 77
Depression (Psychiatric disorders) | 95
Insomnia (Psychiatric disorders) | 135
Cough (Respiratory, thoracic and mediastinal disorders) | 218
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 275
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 136
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 105
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 70
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 88
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 75
Rash (Skin and subcutaneous tissue disorders) | 77

LIMITATIONS AND CAVEATS:
Mean and dispersion for clinical abnormalities were intended to be reported but due to early termination of study (09-Dec-2010) only number and percent of participants are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.